CLINICAL TRIAL: NCT03698500
Title: Blood Level of Specific microRNA Pattern as Potential Biomarker for Inflammatory Bowel Disease
Brief Title: Specific microRNAs as Potential Biomarker for Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FC201603
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-08

CONDITIONS: Crohn's Disease; Ulcerative Colitis
Keywords: Ulcerative Colitis; Crohn's disease; miRNA
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with intestinal colitis and control patients (Other): Device: qPCR diagnostic of specific microRNAs in peripheral blood (10 ml)
  Interventions: Other: Removal of blood

INTERVENTIONS:
Other: Removal of blood — 10 ml of blood will be removed from a peripheral vene during routine diagnostical blood draw

SUMMARY:
The aim of this study is to assess the ability of miR-320a and other specific microRNAs to follow the disease course in patients with Crohn's disease (CD) and ulcerative colitis (UC), and to distinguish both entities, infectious colitis and healthy controls. Furthermore, the accuracy of miRNA-320a to distinguish CD or UC from irritable bowel syndrome (IBS) should be evaluated .

The study is designed as a single center non-randomised prospective trial.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD), which comprises Crohn's disease (CD) and ulcerative colitis (UC), is a chronic-remittent disease of the gastrointestinal tract with leading symptoms such as diarrhea, abdominal pain and rectal bleeding. Absence of mucosal inflammation (so called mucosal healing) is a promising treatment target.as it leads to reduction of colectomy rates, hospitalization and need for surgery. However, overtreatment with severe combined immunosuppressive therapy always bears the risk of severe side-effects such as opportunistic infections. To assess the course of disease, clinical evaluation, noninvasive diagnostic or imaging and invasive endoscopic techniques are currently used. As frequent endoscopical monitoring is not always possible, more specific and noninvasive biomarker are needed to monitor disease activity. The commonly used noninvasive biomarkers C-reactive protein and fecal Calprotectin, which are useful to detect disease activity, are limited due to the lacking specificity for IBD and the weak correlation with the extend of disease. Overall the currently available tools to noninvasively follow the course of disease activity do not possess appropriate specificity, sensitivity and cost effectiveness for in- and outpatient clinical monitoring.

Recently, we could demonstrate the potential of miR(microRNA)-320a to monitor disease activity in experimental colitis mouse models.

The aim of this study is to assess the ability of miR-320a and other specific microRNAs to follow the disease course in patients with inflammatory bowel disease as compared to healthy controls, non IBD-colitis and IBS.

The study is planned as a prospective single center study.

Number of patients: 7 groups of 50 patients

* 1: adult CD patients in remission
* 2: adult CD patient with endoscopical proven disease activity
* 3: adult UC patients in remission
* 4: adult UC patient with endoscopical proven disease activity
* 5: adults with infectious colitis (ie. Ischemic, infectious or toxic colitis)
* 6. Adults with IBS
* 7: healthy adults

All eligible individuals are informed about the nature of the study. All individuals provide written informed consent before entering the trial.

Budget:

All procedures in the present study are performed in ordinary patients, with ordinary staff. Therefore, no extra costs occur for personal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Crohn's disease or ulcerative colitis
* Control patients: healthy patients or patients with colitis of other origin than Crohn's disease or ulcerative colitis as well as patients with IBS

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Inability to understand information for participation
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between microRNA expression level in peripheral blood (qPCR) and disease activity of intestinal Inflammation of CD and UC | 1 day

SECONDARY OUTCOMES:
Assessment of the potential of specific miRNAs to discriminate CD and UC in peripheral blood (qPCR) | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Anna Friederike Cordes, MD, PhD, Principal Investigator — University Hospital Muenster, University of Muenster
Locations (1):
- University of Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No